CLINICAL TRIAL: NCT06075927
Title: An Exploratory Clinical Study of Multivirus-specific T Cells in the Treatment of Refractory Cytomegalovirus and/or Epstein-Barr Virus Infection After Allogeneic Hematopoietic Stem Cell Transplantation
Brief Title: Multivirus-specific T Cells in the Treatment of Refractory CMV and/or EBV Infection After Allo-HSCT
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Peking University People's Hospital (Other)
Responsible Party: Principal Investigator, Xiao-Jun Huang, Professor, Peking University People's Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2023PHD006-001
Record Dates: First submitted 2023-09-12; First posted 2023-10-10 (Actual); Last update posted 2023-10-10 (Actual); Status verified 2023-10

CONDITIONS: CMV Infection; EBV Infection; Stem Cell Transplant
Keywords: Cytomegalovirus; Epstein Barr virus; Multivirus-specific Cytotoxic T-Lymphocytes; Stem Cell Transplant
MeSH Terms: conditions — Cytomegalovirus Infections; Epstein-Barr Virus Infections

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- VSTs infusion (Experimental): Phase I (dose escalation) : An open, single-arm, dose-escalation clinical study to explore the safety, tolerability, and cytodynamic characteristics of CMV and EBV-specific T cells (VSTs), with initial efficacy observations. Subjects enrolled with refractory CMV and/or EBV infection after allogeneic hematopoietic stem cell transplantation were subjected to a 3+3 dose-climb test. Exploring the safety, dose-limiting toxicities (DLT) and maximum tolerated dose (MTD) of intravenous infusion of multi-virus VSTs.
  (2) Phase II (dose expansion) : According to the clinically recommended or safe and effective dose determined by the phase I climb test, the extended study of 1-2 dose groups with 20 cases per dose was performed after joint review by the investigators and project collaborators.
  Interventions: Biological: Virus specific T cells

INTERVENTIONS:
Biological: Virus specific T cells — Subjects will receive partial HLA-matched viral-specific T cells (VSTs) against both CMV and EBV on one of the following dose levels:
  Level One: 1 x 10^7 cells/m2 Level Two: 2 x 10^7cells/m2 Level Three: 5x 10^7 cellss/m2

SUMMARY:
To evaluate the safety and tolerability of partial HLA-matched VSTs against both CMV and EBV viruses in recipients of allogeneic hematopoietic stem cells with refractory viral infections (CMV and/or EBV).

Preliminary evaluation of the efficacy of partial HLA-matched VSTs against both CMV and EBV viruses in recipients of allogeneic hematopoietic stem cells with refractory viral infections (CMV and/or EBV); To monitor the duration and expansion of multi-virus VSTs cells after infusion.

DETAILED DESCRIPTION:
This study consists of two parts: (1) The first stage is the safety evaluation of multi-virus VSTs and the exploration of DLT and MTD; (2) The second phase is to evaluate the safety and efficacy of multi-viral VSTs in selecting appropriate doses in the first phase.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥18 years old, and less than or equal to 70 years old, gender is not limited.
* Prior myeloablative or non-myeloablative allogeneic hematopoietic stem cell transplantation.
* Persistent infection with CMV and/or EBV persists despite standard treatment .
* Prednisone or its equivalent hormone is less than or equal to 0.5 mg/kg/ day when enrolled.
* ECOG score ≤3, expected survival greater than 3 months.
* End blood oxygen saturation ≥90% on room air.
* Available multi-virus-specific cytotoxic T lymphocytes.
* Negative pregnancy test in female patients if applicable.
* Written informed consent and/or signed assent line from patient, parent or guardian.

Exclusion Criteria:

* Within 28 days after allogeneic hematopoietic stem cell transplantation.
* Active III-IV acute GVHD, and/or moderate and above chronic GVHD.
* Severe organ dysfunction: Heart: New York Heart Association (NYHA) levels III and IV; Liver: Total bilirubin>34umol/l; ALT, AST>2 times the normal upper limit; Kidney: Blood creatinine >130umol/L; Lung: Type I or II respiratory failure; Brain: unconsciousness, intracranial hypertension.
* Received DLI, other CTL, CAR-T, NK and other cell therapies, T cell monoclonal antibody immunosuppressants, or participated in any other clinical research related to drugs and medical devices within 28 days before enrollment.
* Poor compliance, and subjects deemed unsuitable for study participation by the investigator.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 29 (Estimated)
Dates: Start 2023-11-01 (Estimated); Primary Completion 2025-07-30 (Estimated); Study Completion 2025-10-30 (Estimated)

PRIMARY OUTCOMES:
Assessment of safety and toxicity outcomes in subjects receiving VSTs infusion | within 56 days after the first VSTs infusion
  Number of participants with treatment-related adverse events as assessed by CTCAE v5.0, and graft-versus-host-disease will be summarized using descriptive statistics for each dose level
Assessment of antiviral efficacy of VSTs infusion | within 56 days after the first VSTs infusion
  Antiviral efficacy including clinical signs of viral infections, virus reinfection, and laboratory measurement of viral load after VSTs infusion will be determined

SECONDARY OUTCOMES:
Virus-specific immune reconstitution | within 56 days after the first VSTs infusion
  Laboratory measurement of virus-specific immune reconstitution before and after VSTs infusion will be tested

CONTACTS AND LOCATIONS:
Overall Officials: Xiangyu Zhao, Study Chair — Peking University People's Hospital

IPD SHARING:
Plan to Share IPD: No